CLINICAL TRIAL: NCT06986681
Title: Effects of Big Toe Muscles Strengthening Exercises With and Without Neuromuscular Training on Speed, Agility and Power Among Runners
Brief Title: Big Toe Muscles Strengthening Exercises With and Without Neuromuscular Training Among Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0453
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sports Physical Therapy
Keywords: Big Toe; Dynamometer; Neuromuscular Training; Runners

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Big toe muscles strengthening exercises (Experimental): 16 Participants will be in experimental group giving them Big toe muscles strengthening exercises protocol along with their normal sports training plan for eight weeks, measuring all values before giving them protocol and after protocol.
  Interventions: Other: Big toe muscles strengthening exercises
- Big toe muscles strengthening exercises with neuromuscular training (Experimental): 16 Participants will be in experimental group giving them Big toe muscles strengthening exercises and neuromuscular training protocol along with their normal sports training plan for eight weeks, measuring all values before giving them protocol and after protocol.
  Interventions: Other: Big toe muscles strengthening exercises with neuromuscular training

INTERVENTIONS:
Other: Big toe muscles strengthening exercises — 16 Participants will be in experimental group giving them Big toe muscles strengthening exercises protocol along with their normal sports training plan for eight weeks, measuring all values before giving them protocol and after protocol
  Arms: Big toe muscles strengthening exercises
Other: Big toe muscles strengthening exercises with neuromuscular training — 16 Participants will be in experimental group giving them Big toe muscles strengthening exercises and neuromuscular training protocol along with their normal sports training plan for eight weeks, measuring all values before giving them protocol and after protocol.
  Arms: Big toe muscles strengthening exercises with neuromuscular training

SUMMARY:
The big toe in relation to the other toes is responsible for a much greater percentage of foot and body stabilization as well as forward propulsion. Big toe muscles play a very significant role in the toe off phase during the locomotion, increasing the final push off from the ground during activities like walking, running and jumping. Also have a role in maintaining medial arch of the foot. Marked evidence shows that neuromuscular training programs are effective for improving measures of performance. Comprehensive neuromuscular training programs designed for young women may significantly increase power, strength, and neuromuscular control. So, this study will determine the effects of big toe muscles strengthening exercises with and without neuromuscular training among runners.

This study will be a randomized clinical trial conducted at Pakistan sports board and coaching center Lahore and runners club in Lahore. Only female runners aged between 18-30 years having at least 1 year experience will be recruited in study. The participants will be randomly divided by simple random sampling into two groups. One group will perform the big toe muscles strengthening exercises with neuromuscular training and the other group will perform the big toe muscles strengthening exercises without neuromuscular training. The effects of Strengthening exercises of both the groups will be accessed on speed, power and agility of runners. Toe strength will be accessed by toe-hip dynamometer, Speed by 30 m sprint test, power by vertical jump, and agility by T-drill agility test at the start, and at the end of study duration. Statistical analysis will be performed using SPSS-26 providing a comprehensive approach to investigate the effects of bio toe muscles strength with and without neuromuscular training on speed, agility and power among runners.

DETAILED DESCRIPTION:
The main objective of the study is to apply the big toe muscles strengthening exercises with and without neuromuscular training and to compare the results to identify their influence on speed, agility and power among runners.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30 years.
* Only female participants.
* Middle distance runners with at least 1 year experience.

Exclusion Criteria:

* Participants with current or recent (< 6 months) lower extremity musculoskeletal symptoms, neurological or neuromuscular conditions, severe foot deformities (i.e. club foot or deformities that hinders the activities of daily living).
* Participants with history of trauma or surgical treatment of lower extremity or foot within 6 months.
* Female participants with pregnancy.
* Systemic illnesses: Diabetes and hypertension etc.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 32 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
30 M sprint test | 8 weeks
  The test involves running a single maximum sprint over 30 meters, with the time recorded. A thorough warm up should be given, including some practice starts and accelerations. Start from a stationary position, with one foot in front of the other. The front foot must be on or behind the starting line. This starting position should be held for 2 seconds prior to starting, and no rocking movements are allowed. The tester should provide hints for maximizing speed (such as keeping low, driving hard with the arms and legs) and encourage them to continue running hard through the finish line. Two trials are allowed, and the best time is recorded to the nearest 2 decimal places. The timing starts from the first movement (if using a stopwatch) or when the timing system is triggered and finishes when the chest crosses the finish line and/or the finishing timing gate is triggered.
T-drill agility test | 8 weeks
  Subjects are asked to sprint forwards 10 yards (9.14 m) from the start line to the first cone and touch the tip with their right hand, shuffle 5yards (4.57 m) left to the second cone and touch with their left hand, then shuffle 10 yards (9.14 m) to the right to the third cone and touch with their right, shuffle 5 yards (4.57 m) back left to the middle cone and touch with their left hand before finally run backwards to the start line. Time began upon subjects passing through the timing gates and stopped upon them passing through on return. The test will not be counted if the subject crosses one foot in front of the other while shuffling, fails to touch the base of the cones, or fails to face forward throughout the test. Take the best time of three successful trials.
Vertical jump test | 8 weeks
  The athlete stands side on to a wall and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked or recorded. This is called the standing reach test. The athlete then stands away from the wall, and leaps vertically as high as possible using both arms and legs to assist in projecting the body upwards. The jumping technique can or cannot use a counter movement. Attempt to touch the wall at the highest point of the jump. The difference in distance between the standing reach height and the jump height is the score. The best of three attempts is recorded.
Toe-Hip Dynamometer | 8 weeks
  The Toe-Hip Strength Dynamometer is a novel IFM dynamometer that has been recently developed for clinicians. Using this tool, the test is conducted similarly to the paper-grip test. This dynamometer is similarly made of a plastic card attached to a hanging scale. For the test, individuals press their toes onto the card as hard as possible without toe curl to resist the assessor pulling the card out, and a peak force output is provided once the card slides out. Although it is still difficult to conclusively isolate the IFM, this device has a lower cost and size compared to other methods and may be useful in clinical settings. Furthermore, the tool is designed for the measurement to occur in a closed-chain position, which is the functional position of the foot.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurihara T, Terada M, Numasawa S, Kusagawa Y, Maeo S, Kanehisa H, Isaka T. Effects of age and sex on association between toe muscular strength and vertical jump performance in adolescent populations. PLoS One. 2021 Dec 31;16(12):e0262100. doi: 10.1371/journal.pone.0262100. eCollection 2021. PMID 34972181
- [Background] Yamauchi J, Koyama K. Importance of toe flexor strength in vertical jump performance. J Biomech. 2020 May 7;104:109719. doi: 10.1016/j.jbiomech.2020.109719. Epub 2020 Feb 26. PMID 32173032
- [Background] Xu J, Goss DD, Saliba SA. A Novel Intrinsic Foot Muscle Strength Dynamometer Demonstrates Moderate-To-Excellent Reliability and Validity. Int J Sports Phys Ther. 2023 Aug 1;18(4):997-1008. doi: 10.26603/001c.84310. eCollection 2023. PMID 37547834
- [Background] Caldemeyer LE, Brown SM, Mulcahey MK. Neuromuscular training for the prevention of ankle sprains in female athletes: a systematic review. Phys Sportsmed. 2020 Nov;48(4):363-369. doi: 10.1080/00913847.2020.1732246. Epub 2020 Feb 28. PMID 32067546
- [Background] Trowell D, Phillips E, Saunders P, Bonacci J. The relationship between performance and biomechanics in middle-distance runners. Sports Biomech. 2021 Dec;20(8):974-984. doi: 10.1080/14763141.2019.1630478. Epub 2019 Jul 31. PMID 31364954
- [Background] Denadai BS, Greco CC. Could middle- and long-distance running performance of well-trained athletes be best predicted by the same aerobic parameters? Curr Res Physiol. 2022 Jun 23;5:265-269. doi: 10.1016/j.crphys.2022.06.006. eCollection 2022. PMID 35800136
- [Background] Kusagawa Y, Kurihara T, Maeo S, Sugiyama T, Kanehisa H, Isaka T. Associations between the size of individual plantar intrinsic and extrinsic foot muscles and toe flexor strength. J Foot Ankle Res. 2022 Mar 21;15(1):22. doi: 10.1186/s13047-022-00532-9. PMID 35313927
- [Background] Willemse L, Wouters EJM, Pisters MF, Vanwanseele B. Plantar intrinsic foot muscle activation during functional exercises compared to isolated foot exercises in younger adults. Physiother Theory Pract. 2024 Aug;40(8):1656-1668. doi: 10.1080/09593985.2023.2204947. Epub 2023 Apr 26. PMID 37126537
- [Background] Rowley M, Kurihara T, Ortiz-Weissberg D, Kulig K. Contributions of flexor hallucis longus and brevis muscles to isometric toe flexor force production. Acta Bioeng Biomech. 2023;25(1):91-99. PMID 38314582
- [Background] van Oeveren BT, de Ruiter CJ, Beek PJ, van Dieen JH. The biomechanics of running and running styles: a synthesis. Sports Biomech. 2024 Apr;23(4):516-554. doi: 10.1080/14763141.2021.1873411. Epub 2021 Mar 4. PMID 33663325